CLINICAL TRIAL: NCT00142428
Title: A Phase II Study of Cetuximab in Patients With Unresectable or Metastatic Hepatocellular Carcinoma
Brief Title: Cetuximab in Patients With Unresectable or Metastatic Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-347
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; cetuximab; Unresectable hepatocellular carcinoma; Metastatic hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental): The initial dose of cetuximab was 400 mg/m2 (cycle 1 only) given intravenously followed by weekly intravenous infusions at 250 mg/m2. Each cycle was defined as 6 consecutive weekly intravenous treatments. Treatment was continued until 1 of the following criteria was met: disease progression per RECIST criteria, unacceptable toxicity, patient refusal, or the need to delay therapy more than 3 weeks.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — The initial dose of cetuximab was 400 mg/m2 (cycle 1 only) given intravenously followed by weekly intravenous infusions at 250 mg/m2. Each cycle was defined as 6 consecutive weekly intravenous treatments. Treatment was continued until 1 of the following criteria was met: disease progression per RECIST criteria, unacceptable toxicity, patient refusal, or the need to delay therapy more than 3 weeks.

SUMMARY:
The main purpose of this study is to begin to collect information and to try to learn whether or not cetuximab works in treating patients with unresectable or metastatic hepatocellular carcinoma.

DETAILED DESCRIPTION:
The first step in this study is to examine the tumor biopsy (previously collected) and determine whether or not it is epidermal growth factor receptor (EGFR) positive or EGFR negative. Both EGFR positive and EGFR negative patients can participate in this study because at this time it is not known whether having a negative or positive receptor makes a difference in how the study drug works on the tumor. By knowing if the tumor is EGFR positive or negative, we will be able to see if there is a difference in the way the tumor responds to cetuximab.

Patients will receive cetuximab intravenously once weekly for 6 weeks. Each 6-week period is one cycle of treatment. The first dose of cetuximab is larger than the following doses.

For the first clinic visit the patient's blood pressure, temperature, breathing and heart rate will be taken before, during, at the end, and one-hour after the cetuximab has been administered. For each visit after that, blood pressure, temperature, breathing and heart rate will be taken before and after cetuximab has been administered.

Before each administration of cetuximab, diphenhydramine will also be administered to decrease the chances of an allergic or hypersensitivity reaction.

The following tests and procedures will be performed at weeks 1, 3 and 5 during each 6-week cycle of treatments as well as at the end of study treatment: physical exam, vital signs, medical history and blood work. At the end of each 6-week cycle a CT and/or MRI will be performed to measure the tumor size.

Long-term follow-up will include physical exams and bloodwork every 6 months.

Patients will remain on cetuximab as long as there is no disease progression or intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic hepatocellular carcinoma
* Measurable tumor
* Adequate hepatic function: total bilirubin < 3.0mg/dl; AST < 7 x upper limit of normal (ULN).
* Adequate renal function: serum creatinine < 2.0mg/dl
* Adequate bone marrow function: absolute neutrophil count (ANC) > 1,000/mm3; platelets > 75,000/mm3.
* 0-2 prior systemic chemotherapy regimens for hepatocellular carcinoma
* 18 years of age and older
* ECOG performance status of 0-2
* Life expectancy > 12 weeks

Exclusion Criteria:

* Surgery, excluding prior diagnostic biopsy or venous access device placement, within 28 days of study entry
* Uncontrolled serious medical or psychiatric illness
* Irradiation or chemotherapy for disease within 28 days of study entry
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Received an investigational agent within 30 days
* Cancer of the Liver Italian Program (CLIP) score > 3
* Acute hepatitis
* Active or uncontrolled infection
* Significant history of cardiac disease
* Prior cetuximab or other therapy which specifically and directly targets the EGFR pathway
* Prior allergic reaction to chimerized or murine monoclonal antibody therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2005-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival in patients treated with cetuximab for unresectable or metastatic hepatocellular carcinoma | 2 years

SECONDARY OUTCOMES:
Number of patients with adverse events | 2 years
Overall Survival | 2 years
Objective Response Rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew X. Zhu, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts